CLINICAL TRIAL: NCT05047887
Title: Comparison of Socket Preservation Using Socket Shield Technique With Autogenous Dentin Graft Versus Alloplast Graft Material (Clinical and Histological Study)
Brief Title: Socket Preservation Using Socket Shield Technique Comparison of Socket Preservation Using Socket Shield Technique With Autogenous Dentin Graft Versus Alloplast Graft Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: socket preservation_2020
Record Dates: First submitted 2021-09-06; First posted 2021-09-17 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Extraction Tooth Socket

STUDY DESIGN:
Intervention Model Description: A single group in a split-mouth design, right and left sides are randomly allocated to the intervention group (16 sides in 8 patients)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (in one side) (Experimental): Modified socket shield technique with autogenous dentin graft
  Interventions: Procedure: Modified socket shield technique with autogenous dentin graft material (in one side)
- Control group (in contrlateral side) (Active Comparator): Modified socket shield technique with alloplast
  Interventions: Procedure: Modified socket shield technique with alloplast graft material (in contralateral side)

INTERVENTIONS:
Procedure: Modified socket shield technique with autogenous dentin graft material (in one side) — The crown of the hopeless tooth will be decoronated, the root will then be sectioned, the lingual root fragment will be carefully retrieved, the remaining buccal root fragment will be thinned and concaved, The coronal part of this shield will be beveled to make a lingual slope then Tooth particles will be demineralized using 2% HNO3 (El-Gomhouria CO. Egypt) for 20 minutes to expose the dentin organic matrix.
  Arms: Study group (in one side)
Procedure: Modified socket shield technique with alloplast graft material (in contralateral side) — The crown of the hopeless tooth will be decoronated, the root will then be sectioned, the lingual root fragment will be carefully retrieved, the remaining buccal root fragment will be thinned and concaved, The coronal part of this shield will be beveled to make a lingual slope then alloplast graft will be used
  Arms: Control group (in contrlateral side)

SUMMARY:
Alveolar bone resorption and labial bone plate reduction follow teeth extraction due to the deficiency of blood supply, derived from the loss of periodontal ligaments, and hence the socket shield technique with autogenous dentine was introduced to preserve the periodontal ligaments.

this study aim to evaluate of socket preservation using alloplast with socket shield versus Autogenous dentin graft with socket shield through radiographic analysis of alveolar bone dimension change and mean bone density in addition to histological and histomorphometric analysis for the quality of the formed bone.

ELIGIBILITY:
Inclusion Criteria:

* One or more of non-restorable (fractured or decayed) tooth/teeth in the maxillary aesthetic regions (incisors, premolars) in both side
* Intact labial periodontal tissues.
* Ability to read and sign an informed consent form.

Exclusion Criteria:

* A medical history that contraindicates oral surgical treatment (uncontrolled/untreated diabetes mellitus, immunocompromised status, radio/chemotherapy of the oral and maxillofacial region, treatment with oral and/or intravenous amino-bisphosponates).
* Untreated periodontal disease.
* Vertical root fractures on the labial aspect.
* Tooth /teeth with horizontal fractures below bone level.
* Tooth /teeth with external or internal resorptions.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
post opertaive edema | after 7 days
  This will be assessed in the 1st week postoperatively and measured as follows: None (no inflammation) Mild (intraoral swelling confined to the surgical field) Moderate (extraoral swelling in the surgical zone) Severe (extraoral swelling spreading beyond the surgical zone).
change in pain score | 1 week and 3 months
  it will be assessed using VAS It rates pain on a scale from 1-10, with 0 representing "no pain" and 10 "very much pain
Change in bone density | at baseline and 3 months
  it will be assessed using CBCT
Change in bone height | at baseline and 3 months
  it will be assessed using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt